CLINICAL TRIAL: NCT02471183
Title: Multicenter, Open-label, Single-group Study to Assess the Tolerability and the Safety of the Transition From Inhaled Treprostinil to Oral Selexipag in Adult Patients With Pulmonary Arterial Hypertension
Brief Title: Study to Assess the Tolerability and the Safety of the Transition From Inhaled Treprostinil to Oral Selexipag in Patients With Pulmonary Arterial Hypertension
Acronym: TRANSIT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-065A304
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Results first posted 2017-12-28 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — selexipag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selexipag, Open Label (Experimental): Subjects on inhaled treprostinil treatment participate in a 16-week main treatment period including down-titration of treprostinil to end of Week 8 and parallel up-titration of selexipag to the maximum tolerated dose (MTD) up to Week 12, for each individual patient but not above 1600 mcg twice daily.
  From Week 12 up to Week 16, patients continue selexipag at their individual MTD. Patients could continue the study drug selexipag during the extended treatment period from Week 16 until commercial availability of selexipag.
  Interventions: Drug: Selexipag

INTERVENTIONS:
Drug: Selexipag — Tablets for oral administration containing 200 micrograms (mcg) of selexipag to be administered twice a day. The individual dose is to be established during the first 12 weeks of the study. Doses are in the range from 200 micrograms (1 tablet) to 1,600 micrograms (8 tablets).
  Other Names: Uptravi; ACT-293987

SUMMARY:
This study enrolls patients with pulmonary arterial hypertension (PAH) treated with inhaled treprostinil. During the study, the treatment with inhaled treprostinil will be tapered off and simultaneously replaced with an oral treatment (selexipag) targeting the disease in a similar way. The purpose of the study is i) to investigate the safety and tolerability of oral selexipag in patients who transition from inhaled treprostinil, ii) to investigate the effects of oral selexipag on PAH severity and exercise ability before and after transition, and iii) to gain new information about the patients experience taking oral selexipag compared to inhaled treprostinil. Study participants may stay in the study until the FDA has granted marketing authorization.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged from 18 to 75 years (inclusive) with pulmonary arterial hypertension (PAH).
* Etiology of PAH belonging to one of the following subgroups: idiopathic PAH, Heritable PAH, drug or toxin induced, associated with connective tissue disease, associated with HIV infection, associated with congenital heart disease with simple systemic-to-pulmonary shunt at least 1 year after surgical repair.
* Women of childbearing potential are eligible only if the following apply: Negative serum pregnancy test at Visit 1 and a negative urine pregnancy test at Visit on Day 1, agreement to undertake monthly urine pregnancy tests during the study and up to 30 days after study drug discontinuation, agreement to use efficient methods of birth control from Visit 1 up to at least 30 days after study treatment discontinuation.
* Documented hemodynamic diagnosis of PAH by right heart catheterization (RHC).
* Inhaled treprostinil treatment ongoing for at least 90 days and at stable dose for at least 30 days prior to Day 1.
* WHO functional class (FC) II or III at Visit 1 and Visit 2.
* 6-minute walk distance (6MWD) ≥ 300 m at Visit 1.
* On background oral PAH therapy for at least 90 days and on a stable dose for 30 days prior to Visit 2. Acceptable concomitant PAH therapies are one or two of the following: a) Endothelin receptor antagonist (ERA), b) Phosphodiesterase type 5 (PDE-5) inhibitor or soluble guanylate cyclase (sGC) stimulator.

Exclusion Criteria:

* Treatment with any prostacyclin or prostacyclin analogs other than inhaled treprostinil within 90 days before Day 1, or patients scheduled to receive any of these treatments within the duration of the study.
* Any hospitalization within 90 days before Day 1.
* Worsening in WHO FC within 30 days prior to Day 1.
* At any time prior to Day 1, documented moderate or severe obstructive or restrictive lung disease.
* Known or suspicion of pulmonary veno-occlusive disease (PVOD).
* Anemia: < 80 g/L (5.0 mmol/L) hemoglobin.
* Clinically relevant thyroid disease (hypo- or hyperthyroidism).
* Known and documented severe hepatic impairment.
* Uncontrolled hypertension.
* Sitting systolic blood pressure < 85 mmHg.
* Acute myocardial infarction within the last 90 days prior to Visit 1.
* History of left-sided heart disease.
* Left ventricular disease/dysfunction risk factors.
* Documented pericardial effusion within 90 days prior to Visit 1.
* Documented severe renal insufficiency.
* Receiving or having received any investigational drugs within 90 days before Day 1.
* Having received selexipag at any time before Day 1.
* Acute or chronic impairment (other than dyspnea), limiting the ability to comply with study requirements.
* Recently conducted or planned cardio-pulmonary rehabilitation program based on exercise training during the study.
* Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements.
* Known concomitant life-threatening disease with a life expectancy < 12 months.
* Females who are lactating or pregnant or plan to become pregnant during the study.
* Known hypersensitivity to any of the excipients of the drug formulation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2016-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - UCSD Medical Center -La Jolla, La Jolla, California
  - UCSF Medical Center, San Francisco, California
  - Harbor UCLA Medical Center, Torrance, California
  - Emory University, Atlanta, Georgia
  - Piedmont Healthcare Research Institute, Austell, Georgia
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Duke Unversity, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Sentara Cardiovascular Research Instistute, Norfolk, Virginia

REFERENCES:
- [Derived] Frost A, Janmohamed M, Fritz JS, McConnell JW, Poch D, Fortin TA, Miller CE, Chin KM, Fisher M, Eggert M, McEvoy C, Benza RL, Farber HW, Kim NH, Pfister T, Shiraga Y, McLaughlin V. Safety and tolerability of transition from inhaled treprostinil to oral selexipag in pulmonary arterial hypertension: Results from the TRANSIT-1 study. J Heart Lung Transplant. 2019 Jan;38(1):43-50. doi: 10.1016/j.healun.2018.09.003. Epub 2018 Sep 12. PMID 30391194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-seven patients were screened. Among them, thirty-four patients with pulmonary arterial hypertension (PAH) and treated with inhaled treprostinil for at least 90 days were enrolled at 12 sites in the USA.
Groups:
- Selexipag: The subjects participated in a 16-week main treatment period including down-titration of treprostinil to end of Week 8 and parallel up-titration of selexipag to the maximum tolerated dose (MTD) up to Week 12, for each individual patient but not above 1600 mcg twice daily.
  From Week 12 up to Week 16, patients continued selexipag at their individual MTD. Patients could continue the study drug selexipag during the extended treatment period from Week 16 until commercial availability of selexipag.
Period: Main Treatment Period
Arm/Group | Selexipag
Started | 34
Completed | 32
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Extended Treatment Period
Arm/Group | Selexipag
Started | 32
Completed | 31
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Selexipag
Number analyzed (Participants) | 34
Age, Customized [Count of Participants; unit: Participants]
  Age categories as per protocol: <= 65 years | 28
  Age categories as per protocol: >65 years and <75 years | 5
  Age categories as per protocol: >= 75 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race categories as per protocol: Black or African American | 2
  Race categories as per protocol: Asian | 3
  Race categories as per protocol: White | 28
  Race categories as per protocol: Other | 1
Etiology of pulmonary arterial hypertension (PAH) [Count of Participants; unit: Participants] — Patients included in the study had a diagnosis of PAH belonging to one of the following categories at screening:
  * Idiopathic PAH
  * Heritable PAH
  * Drug or toxin induced PAH
  * PAH associated with connective tissue disease or HIV infection or congenital heart disease
  Participants
    Idiopathic | 19
    Heritable | 0
    Drug or toxin induced | 5
    Associated PAH | 10
World Health Organization Functional class (WHO FC) [Count of Participants; unit: Participants] — The World Health Organization (WHO) defines 4 classes to classify the functional status of patients with pulmonary hypertension:
  Class I (FC I): No limitation of physical activity; Class II (FC II): Slight limitation of physical activity; Class IIII (FC III): Marked limitation of physical activity; Class IV (FC IV): Inability to carry out any physical activity without symptoms.
  Number of subjects in each WHO FC category before the first study drug administration is reported here.
  Participants
    FC I | 0
    FC II | 25
    FC III | 9
    FC IV | 0
Time since initial inhaled treprostinil [Median (Full Range); unit: Months] — This is the time elapsed since initiation of treatment with inhaled treprostinil and before starting the study drug selexipag.
  Months | 37.8 [4.4 to 135.2]
Treprostinil stable dose [Count of Participants; unit: Participants] — This corresponds to the daily stable dose of inhaled treprostinil before initiation of selexipag based on the prescribed dose within 30 days before the intiation of selexipag (Day 1). The stable dose of treprostinil is expressed in mcg q.i.d., which is the number of breaths per 4 treatment session per day x 6 mcg
  Participants
    < 54 mcg q.i.d. | 2
    54 mcg q.i.d. | 20
    > 54 mcg q.i.d. | 12
PAH-specific therapy at baseline [Count of Participants; unit: Participants] — Number of patients receiving any of the following oral PAH background medication for at least 90 days prior to study treatment with selexipag:
  Endothelin Receptor Antagonists (ERAs) or Phosphodiesterase-5 (PDE5) inhibitor or Soluble guanylate cyclase (sGC) stimulator or a combination of these therapeutic classes
  Participants
    PDE5-inhibitors alone | 7
    ERAs alone | 4
    ERAs and PDE-5 | 19
    ERAs and sCG stimulator | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Sustained Treatment Transition
Description: A sustained treatment transition is considered if the 3 following criteria are met a) being on study treatment (selexipag) at Week 16, and b) not having a study treatment interruption(s) of a total of 8 days or more prior to Week 16, and c) absence of inhaled treprostinil or any prostanoid treatment after Week 8 up to Week 16.
  The percentage of subjects with a sustained treatment transition is calculated with 95% confidence interval (CI) using the Clopper-Pearson method.
Time Frame: At Week 16
Population: All subjects who took at least one dose of selexipag were included in the safety analyses
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selexipag
Number analyzed (Participants) | 34
Percentage of participants | 82.4 [65.5 to 93.2]

2. Primary Outcome: Percentage of Subjects With Treatment-emergent Adverse Events (AEs),
Description: Percentage of subjects with treatment-emergent AEs (serious and non serious), regardless of relationship to selexipag
Time Frame: 26 weeks on average (from the first dose of selexipag up to 30 days after the last dose of selexipag)
Population: All subjects who took at least one dose of selexipag were included in the safety analyses
Measure: Number; unit: Percentage of participants
Arm/Group | Selexipag
Number analyzed (Participants) | 34
Percentage of participants | 97.1

3. Primary Outcome: Number of Subjects With Adverse Events Leading to Premature Discontinuation of Selexipag
Description: Number of subjects with adverse events leading to premature discontinuation of selexipag is determined from the first dose of selexipag up to the last dose of selexipag
Time Frame: Up to 22 weeks on average
Population: All subjects who took at least one dose of selexipag were included in the safety analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 34
Participants | 3

4. Primary Outcome: Absolute Change From Baseline Over Time in Blood Pressure
Description: Both systolic(SBP) and diastolic (DBP) arterial blood pressure were measured in a sitting position after at least 5 minutes of rest at scheduled time points. Median change from baseline to pre-specified post-baseline visits are calculated
Time Frame: Baseline, Week 4, Week 12, Week 16
Population: All subjects who took at least one dose of selexipag were included in the safety analyses
Measure: Median (Full Range); unit: mmHg
Arm/Group | Selexipag
Number analyzed (Participants) | 34
mmHg
  SBP change from baseline at week 4 | 1.00 [-32.0 to 59.0]
  SBP change from baseline at week 12 | -3.00 [-28.0 to 35.0]
  SBP change from baseline at week 16 | -4.00 [-24.0 to 25.0]
  DBP change from baseline at week 4 | -3.00 [-26.0 to 34.0]
  DBP change from baseline at week 12 | -4.00 [-30.0 to 48.0]
  DBP change from baseline at week 16 | -6.00 [-21.0 to 15.0]

5. Primary Outcome: Absolute Change From Baseline Over Time in Heart Rate (HR)
Description: Pulse rate is measured after at least 5 minutes of rest in a sitting position. Median change from baseline to pre-specified post-baseline visits are calculated.
Time Frame: Baseline, Week 4, Week 12, Week 16
Population: All subjects who took at least one dose of selexipag were included in the safety analyses
Measure: Median (Full Range); unit: beats per minute (bpm)
Arm/Group | Selexipag
Number analyzed (Participants) | 34
beats per minute (bpm)
  HR change from baseline at week 4 | 4.00 [-23.0 to 22.0]
  HR change from baseline at week 12 | 6.00 [-34.0 to 33.0]
  HR change from baseline at week 16 | 3.00 [-35.0 to 23.0]

6. Primary Outcome: Maximal Tolerated Dose
Description: This is the individual maximal tolerated dose (MTD) observed at Week 12 in the subjects still on selexipag at Week 16.
  MTD is defined as the dose of selexipag reached with the last dose change up to Week 12
Time Frame: At Week 12, in subjects still on selexipag at Week 16
Population: Sensitivity analysis: only patients being on selexipag at week 16 are considered.
Measure: Median (Full Range); unit: mcg
Arm/Group | Selexipag
Number analyzed (Participants) | 32
mcg | 1200 [400 to 1600]

7. Primary Outcome: Time to Discontinuation of Inhaled Treprostinil.
Description: Median time from baseline (Day1) to the end of down-titration of inhaled treprostinil is calculated
Time Frame: Baseline to Week 16
Population: All subjects who took at least one dose of selexipag were included in the safety analyses
Measure: Median (Full Range); unit: weeks
Arm/Group | Selexipag
Number analyzed (Participants) | 34
weeks | 6.21 [1.0 to 14.9]

8. Secondary Outcome: Percentage of Subjects With WHO Functional Class (FC) Change From Baseline
Description: The World Health Organization (WHO) defines 4 classes to classify the functional status of patients with pulmonary hypertension:
  Class I (FC I): No limitation of physical activity. Class II (FC II): Slight limitation of physical activity. Class III (FC III): Marked limitation of physical activity. Class IV (FC IV): Inability to carry out any physical activity without symptoms.
  Number of patients with improvement (shift from a higher to a lower class), worsening (shift from a lower to a higher class) or no change in WHO functional class at end of study compared to baseline are determined.
Time Frame: Baseline and Week 16
Measure: Number; unit: percentage of participants
Arm/Group | Selexipag
Number analyzed (Participants) | 34
percentage of participants
  % subjects with WHO FC improvement | 26.5
  % subjects with WHO FC worsening | 5.9
  % subjects with WHO FC unchanged | 67.6

9. Secondary Outcome: Absolute Change in 6-minute Walk Distance (6MWD) at Trough
Description: The 6MWT is a non-encouraged test, which measures the distance (in meters) covered by the subject during a 6-minute walk. It is performed in a 30-meters long flat corridor, where the patient is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed.
  Absolute change from baseline to Week 16 in 6MWD is measured at trough levels of inhaled treprostinil and/or selexipag. The trough level of inhaled treprostinil is defined as the last dose having been taken not less than 4 hours and not more than 48 hours prior to the 6MWT at Visit 1 (screening). The trough level of selexipag was defined as the last dose having been taken not less than 8 hours and not more than 7 days prior to the 6MWT at Visit 5 (Week 16).
Time Frame: Baseline and Week 16
Measure: Median (95% Confidence Interval); unit: meters
Arm/Group | Selexipag
Number analyzed (Participants) | 34
meters | -10.25 [-25.60 to 8.80]

10. Secondary Outcome: Percentage of Patients With Change in 6-minute Walk Distance (6MWD)
Description: Percentage of patients with an increase (> 8% of baseline), maintenance (+/- 8% of baseline), or decrease (< -8% of baseline) in their 6MWD (at trough) from baseline to Week 16. The ± 8% boundaries for change in 6MWD reflect the approximately 8% coefficient of variation in the reproducibility of the 6MWD.
  The trough level of inhaled treprostinil is defined as the last dose having been taken not less than 4 hours and not more than 48 hours prior to the 6MWD test at Visit 1 (screening). The trough level of selexipag was defined as the last dose having been taken not less than 8 hours and not more than 7 days prior to the 6MWD test at Visit 5 (Week 16).
Time Frame: Baseline and Week 16
Measure: Number; unit: Percentage of participants
Arm/Group | Selexipag
Number analyzed (Participants) | 34
Percentage of participants
  6MWD decreased | 26.5
  6MWD maintained | 55.9
  6MWD increased | 17.6

11. Secondary Outcome: Geometric Mean of the Ratio in N-terminal Pro B-type Natriuretic Peptide (NT-proBNP) of Week 16 to Baseline
Description: Changes in NT-proBNP levels in plasma are expressed by the geometric mean of the ratio of Week 16 to baseline
Time Frame: Baseline and Week 16
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean of the ratio
Arm/Group | Selexipag
Number analyzed (Participants) | 34
Geometric mean of the ratio | 1.1 [0.82 to 1.62]

12. Other Pre Specified Outcome: Change From Baseline to Week 16 in the Treatment Satisfaction Questionnaire for Medication Questionnaire (TSQM II)
Description: The Treatment Satisfaction Questionnaire for Medication, Version II (TSQM II) is a validated tool that evaluate the subject's satisfaction with the study treatment. It includes a total of 11 questions related to satisfaction with treatment effectiveness, side effects,convenience, and global satisfaction.
  TSQM scores range from 0 to 100 for each domain; a higher score indicates higher satisfaction with treatment.
Time Frame: Baseline and Week 16
Measure: Median (95% Confidence Interval); unit: Units on a scale
Arm/Group | Selexipag
Number analyzed (Participants) | 34
Units on a scale
  Effectiveness (change from baseline) | 0.00 [-8.3 to 8.3]
  Side effects (change from baseline) | 0.00 [-16.7 to 0.0]
  Convenience (change from baseline) | 44.44 [27.8 to 61.1]
  Global satisfaction (change from baseline) | 8.33 [0.0 to 25.0]

ADVERSE EVENTS:
Time Frame: From study treatment initiation up to 30 days after study treatment discontinuation
Groups:
- Selexipag: All subjects who take at least one dose of selexipag. The mean duration of exposure to selexipag was 21.6 weeks
Arm/Group | Selexipag
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 2/34
Other Adverse Events (participants affected / at risk) | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selexipag (N=34)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selexipag (N=34)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Brain natriuretic peptide increased (Investigations) | 3 (3)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 24 (32)
Dizziness (Nervous system disorders) | 7 (10)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Fatigue (General disorders) | 8 (10)
Flushing (Vascular disorders) | 8 (11)
Headache (Nervous system disorders) | 27 (40)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (11)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (7)
Oedema peripheral (General disorders) | 5 (6)
Pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 16 (18)
Paraesthesia (Nervous system disorders) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Presyncope (Nervous system disorders) | 3 (4)
Pyrexia (General disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation.

Upon review, Actelion may provide comments, and may also request changes for the sole purpose of protecting its confidential information and/or patent rights.

Neither the institution nor the investigator should permit publication during such a review period.